CLINICAL TRIAL: NCT04217291
Title: Evaluation of the Efficacy and Safety of Different Doses of SY-004 in Patients With Type 2 Diabetes Mellitus
Brief Title: The Efficacy and Safety of Different Doses of SY-004 in Patients With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Suzhou Yabao Pharmaceutical R&D Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SY004003
Record Dates: First submitted 2019-12-30; First posted 2020-01-03 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2021-05

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- SY-004-1 (Experimental): a dose of 80mg/day taken orally for two weeks, and a dose of 80mg/day for 14 weeks from the third week
  Interventions: Drug: SY-004
- SY-004-2 (Experimental): a dose of 80mg/day taken orally for two weeks, and a dose of 160mg/day for 14 weeks from the third week.
  Interventions: Drug: SY-004
- SY-004-3 (Experimental): a dose of 80mg/day orally in the first week, a dose of 160mg/day in the second week and a dose of 240mg/day for 14 weeks from the third week.
  Interventions: Drug: SY-004
- placebo (Placebo Comparator): a dose of SY-004 matching placebo taken orally
  Interventions: Other: SY-004 matching placebo

INTERVENTIONS:
Drug: SY-004 — Take orally once a day
  Arms: SY-004-1; SY-004-2; SY-004-3
Other: SY-004 matching placebo — Take orally once a day
  Arms: placebo

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled phase II clinical study in patients with type 2 diabetes mellitus (T2DM).

DETAILED DESCRIPTION:
200 cases will be included and divided into four groups with 50 cases in each group

ELIGIBILITY:
Inclusion Criteria:

* Gender is not limited.
* Age at screening: ≥ 18 years old, ≥ 75 years old.
* According to WHO diagnostic criteria and classification in 1999, type 2 diabetes was diagnosed, with a course of at least 3 months.
* During screening and before randomization, 18kg / m2 ≤ BMI ≤ 35kg / m2.
* At the time of screening, they had been treated with diet or exercise for at least 3 months.
* No antidiabetic drugs were used at the time of screening, or the antidiabetic drugs were used irregularly within 3 months before screening (the cumulative use of antidiabetic drugs in the past 3 months was no more than 2 weeks and no antidiabetic drugs were used in the past 1 month).
* During screening, 7% of the samples detected by local laboratory were ≤ HbA1c ≤ 11%.
* Before randomization, the central laboratory tested 7% ≤ HbA1c ≤ 11%.
* Fasting blood glucose (FBG) of 7-13.3 mmol / L (including boundary value) was measured in the central laboratory before randomization.
* The subjects must have informed consent before the study, and signed the written informed consent voluntarily.
* The subjects were willing and able to use the home blood glucose meter for self blood glucose monitoring.
* The subjects were able to communicate well with the researchers and complete the study according to the protocol.

Exclusion Criteria:

* Staff members and their immediate family members of the research project. Lineal relatives refer to persons with consanguineous or legal relationships, including spouses, parents, children, brothers and sisters.
* Any of the following drugs or treatments were used prior to screening:

  1. In the past six months, insulin therapy has been used for more than one month, or insulin therapy is needed at present.
  2. Long acting GLP-1 has been used in the past 6 months.
  3. Glucokinase activator (GKA) was used in the past 6 months.
  4. In the past 6 months, I have received weight-loss drugs or any weight-loss treatment (such as surgery, excessive diet and exercise therapy) that leads to weight instability.
  5. Participated in clinical trials of any drug or medical device in the past 3 months.
  6. Other drugs that may affect blood glucose metabolism have been used in the past 8 weeks, including growth hormone treatment, and long-term or repeated intermittent systemic glucocorticoids (intravenous, oral or intra-articular administration for more than 2 weeks or repeated courses, except inhalation or local external use), etc.
  7. Strong CYP3A inducers or strong CYP3A inhibitors have been used in the past two weeks or are planned to be used in the near future (refer to appendix 12.5.1).
  8. Drugs that are likely to cause torsade de pointes have been used in the past two weeks or planned in the near future (refer to appendix 12.5.2).
* Prior to screening, there was a history or evidence of any of the following diseases:

  1. Type 1 diabetes, special type diabetes and secondary diabetes.
  2. Significant clinical cardiovascular events have occurred in the past 6 months (refer to appendix 12.3).
  3. Patients with clinically significant peripheral vascular lesions, such as ischemic ulcer or gangrene, diabetic foot ulcer and infection.
  4. There is sufficient evidence for the presence of active diabetic proliferative retinopathy or maculopathy that is unstable or in need of treatment.
  5. there are obvious autonomic neuropathy, such as urinary retention, orthostatic hypotension, diabetic diarrhea or gastroparesis.
  6. Have a history of acute or chronic pancreatitis.
  7. Ketoacidosis, diabetic acidosis or hyperosmolar nonketotic coma have occurred in the past 6 months and need to be hospitalized.
  8. In the past 6 months, serious hypoglycemic events with unknown causes (need other people's help to recover); or frequent hypoglycemia: for example, more than two hypoglycemic events (blood glucose ≤ 3.9mmol / L) occurred in the first month before screening.
  9. Any endocrine system disease related to blood glucose (such as hyperthyroidism, acromegaly, Cushing's syndrome), immune system disease or other diseases that are unstable or need treatment are not suitable for the study according to the judgment of researchers.
  10. Have other diseases that affect glucose metabolism or are taking drugs that significantly affect glucose metabolism.
  11. Severe trauma or acute infection that may affect blood glucose control has occurred in the past month.
  12. Suffer from serious cardiovascular disease, respiratory system disease, gastrointestinal disease, liver dysfunction, renal dysfunction, endocrine disease (except diabetes), blood system disease, nervous system disease, and the disease status can significantly change the absorption, distribution, metabolism and excretion of the test drug, or taking the test drug will increase the risk of the subject or affect the analysis of the research results.
  13. There are any types of malignant tumors (whether cured or not).
  14. A history of diseases that may cause hemolysis or red blood cell instability that affect HbA1c detection, such as hemoglobinopathy (such as sickle cell anemia or thalassemia, ferriblastic anemia).
  15. History of alcohol and drug abuse. Drink more than 21 units (male) or 14 units (female) of alcohol per week (1 unit is about 360 ml of beer or 45 ml of spirits or 150 ml of wine with 40% alcohol).
  16. There are mental or nervous system diseases, unwillingness to communicate or language barriers, and insufficient understanding and cooperation.
* There is any laboratory inspection index meeting the following standards at screening or random:

  1. In the absence of pacemaker, 12 lead ECG showed second or third degree atrioventricular block, or corrected qtcb > 450ms (male) or > 470ms (female).
  2. eGFR<60ml/(min•1.73m2)。
  3. ALT > 1.5 times the upper limit of normal value (× ULN), AST > 1.5 × ULN, TBIL > 1.5 × ULN.
  4. Hypertension (systolic blood pressure ≥ 160mmhg or diastolic blood pressure ≥ 100mmhg) that cannot be controlled by drugs or other treatment means exists.
  5. Hypertriglyceridemia (triglyceride > 500mg / dl (5.70mmol / L)) was found which could not be controlled by drugs or other treatments.
  6. Hemoglobin < 90g / L.
  7. The serological evidence of infectious virus is positive, including hepatitis B, hepatitis C, HIV and Treponema pallidum.
  8. Fasting C-peptide < 1.0 ng / ml (333 pmol / L).
* Fertile eligible subjects (men and women) disagreed with the use of reliable contraceptive methods during the study and at least one month after the last administration.
* Pregnant or lactating women.
* Allergic to the active ingredient agratine hydrochloride, or severe allergic constitution / severe allergic history.
* Other circumstances judged by the sponsor or researcher as unsuitable for the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2019-12-10 (Actual); Primary Completion 2021-07-09 (Actual); Study Completion 2021-07-09 (Actual)

PRIMARY OUTCOMES:
Changes in Glycosylated Hemoglobin A1c (HbA1c) | 16 weeks
  Changes in Glycosylated Hemoglobin A1c relative to baseline at 16 weeks compared to placebo.

SECONDARY OUTCOMES:
the proportion of subjects whose Glycosylated Hemoglobin A1c (HbA1c) was less than 7%. | 16 weeks
  At the end of 16 weeks, the proportion of subjects whose Glycosylated Hemoglobin A1c was less than 7% .
The proportion of subjects with Glycosylated Hemoglobin A1c (HbA1c) < 6.5% | 16 weeks
  The proportion of subjects with Glycosylated Hemoglobin A1c < 6.5% at 16 weeks after administration of SY-004.
Changes in Glycosylated Hemoglobin A1c (HbA1c) | 8 weeks
  The change of Glycosylated Hemoglobin A1c relative to the baseline after 8 weeks of treatment with SY-004.
the proportion of subjects whose Glycosylated Hemoglobin A1c (HbA1c) was less than 7% | 8 weeks
  At the end of 8 weeks, the proportion of subjects whose Glycosylated Hemoglobin A1c was less than 7% .
The proportion of subjects with Glycosylated Hemoglobin A1c (HbA1c) < 6.5% | 8 weeks
  The proportion of subjects with Glycosylated Hemoglobin A1c < 6.5% at the end of 8 weeks.
Changes in fasting blood glucose (FPG) relative to the baseline | 1、2、4、8、12、16weeks
  Changes in fasting blood glucose (FPG) relative to the baseline at 1, 2, 4, 8, 12 and 16 weeks after administration of SY-004.
Changes in postprandial blood glucose auc0-2h | 16 weeks
  Changes in postprandial blood glucose auc0-2h ( 0-2h blood glucose AUC of Mixed-Meal-Tolerance-Test ) relative to baseline at 16 weeks after administration of SY-004.
Changes in abdominal weight relative to baseline at 8 and 16 weeks. | 8、16weeks
  Changes in abdominal weight relative to baseline at 8 and 16 weeks after administration of SY-004.

CONTACTS AND LOCATIONS:
Overall Officials: Mu, Principal Investigator — Chinese PLA General Hospital
Locations (1):
- PLA General Hospital, Beijing, Beijing Municipality, China